CLINICAL TRIAL: NCT06101589
Title: Effect of Vitamin D Supplementation on the Allostatic Load and Chronic Stress Along Line of Control in Azad Jammu and Kashmir. "Double Blind Randomized Placebo-controlled Trial"
Brief Title: Effect of Vitamin D Supplementation on Allostatic Load and Chronic Stress Along Line of Control in Azad Jammu Kashmir
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Punjab (Other)
Responsible Party: Principal Investigator, Jawwad Afzal Kayani, principal investigator, University of the Punjab
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: D/142/FIMS
Record Dates: First submitted 2023-10-12; First posted 2023-10-26 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Mental Health Issue
MeSH Terms: interventions — Vitamin D; Calcifediol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm in which we will give the active Vitamin D to participants (Experimental): the intervention will be the Vitamin D in its active form 200,00 IU 25(OH)D3.route of administration is oral.
  Interventions: Dietary Supplement: 25 hydroxy cholecalciferol (Vitamin D) /25(OH)D3.
- placebo arm in which we will give the placebo (Placebo Comparator): olive oil will be the placebo medicine. the placebo medicine have similar taste and quantity. the route of administration is oral.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 25 hydroxy cholecalciferol (Vitamin D) /25(OH)D3. — 5 mg (200,000 IU) vitamin D3 in 1 ml ethyl oleate Pharmaceutical form: Solution of vitamin D3 in ethyl oleate, 0.75% w/v. three doses will be given orally every a month apart.
  Arms: experimental arm in which we will give the active Vitamin D to participants
Dietary Supplement: Placebo — Olive oil in 1 ml ethyl oleate with no vitamin D3 content
  Arms: placebo arm in which we will give the placebo

SUMMARY:
FULL TITLE Effect of vitamin D supplementation on the Allostatic load and Chronic stress along line of control in Azad Jammu and Kashmir. "Double blind randomized placebo-controlled trial"

SHORT TITLE Effect of vitamin D supplementation on allostatic load and chronic stress along line of control in azad Jammu and Kashmir PROTOCOL/VERSION DATE 5th August 2023 METHODOLOGY "Double blind randomized placebo-controlled trial"

STUDY DURATION 1 year STUDY CENTRES 1. District head quarter hospital haveli district Azad Kashmir 2. Rural health center (RHC) Khursheed Abad, 3. Basic health unit (BHU) Kirni Mandhaar and 4. First aid post (FAP) Chirikot. Main Objectives -To determine whether high-dose oral vitamin D supplementation effects allostatic load and chronic stress of the residents of line of control haveli district Azad Jammu and Kashmir (primary outcome)

* To assess the prevalence and determinants of allostatic load and chronic stress among the residents of line of control (secondary outcome factors analysis).
* To look into the relationship between chronic stress and vital clinical markers as blood pressure, BMI, and lipid profile in participants from line of control.
* To determine whether this intervention is safe and well-tolerated by study participants (secondary outcomes, safety) No. of Participants 120 Statistical Methodology and Analysis The collected data will be analysed using appropriate statistical techniques: Descriptive statistics will summarize participant characteristics, chronic stress, psychological well-being, physical health indicators, and baseline vitamin D levels. Inferential statistics, such as t-tests, ANOVA, and regression analysis, will be used to examine relationships between chronic stress, allostatic load, vitamin D supplementation, and health outcomes. Subgroup analyses will explore potential interactions based on demographic variables

DETAILED DESCRIPTION:
The aim of this research is to fully comprehend the complex relationship between chronic stress, physiological dysregulation (as measured by allostatic load), and the potential impact of vitamin D supplementation on psychological well-being and physical health in a conflict-affected population.TRIAL ENDPOINTS Primary endpoint The primary outcome will be the Allostatic load after the 3 supplementation doses of study medication.

Secondary Efficacy Endpoints Serum concentration of vitamin D, HbA1C, lipid profile (HDL and LDL), serum cortisol and C reactive proteins after 4 months.

Any change in the Biophysical parameters (blood pressure (BP), heart rate (HR), body mass index (BMI) and hip waist ratio (HRR) after 4 months Chronic stress reduction after 4 months (dose effect) and determinants identification by sub group analysis.

Residents of warzone areas, such as District Haveli in Azad Kashmir, endure persistent exposure to chronic stressors resulting from conflict-related violence, displacement, and traumatic events. This chronic stress not only takes a toll on their mental health but also triggers physiological dysregulation across multiple systems, contributing to an increased allostatic load. Furthermore, the prevalent deficiency of vitamin D, exacerbated by limited sunlight exposure and disrupted food supplies, poses additional health risks in this population. Despite these challenges, there is a notable lack of comprehensive research investigating the determinants of allostatic load in the context of chronic stress and the potential ameliorative effects of vitamin D supplementation. Addressing this gap is crucial for understanding the intricate interplay between stress, physiological health, and potential interventions, thereby contributing to the well-being and resilience of residents in conflict-affected regions.STUDY DESIGN/STUDY PLACE:

The study will employ a It will be a double blinded, parallel individually randomized control trial and will be conducted in District Haveli, Azad Kashmir, armed conflicted area affected by conflict-related stressors.

STUDY POPULATION:

The study will include adult male/female) age (18-60 years) residents of District Haveli, Azad Kashmir, who have been exposed to war-related stressors, violence, and displacement.

SAMPLE SIZE Assuming that 60% of the participants in the control group arm would attain >30% of the baseline vitamin D status at 6 months, we calculated that a total of 94 participants (47 per arm) would need to complete follow-up in order to detect a 25% absolute increase (to 85%) in the proportion of patients attaining >30% vitamin D level at 6 months in the intervention arm with 80% power at the5% significance level(Giacomet et al., 2014). This number will be inflated to a total of 114 allow attrition due to death and loss to follow up. There will be interim analysis in the plan.

SAMPLING TECHNIQUE: The multi-stage cluster sample strategy is ideal for research done in places with geographical dispersion, limited access, and community-specific characteristics. STUDY TOOL:

The study will utilize a combination of validated questionnaires and physiological measurements to collect data.

DATA COLLECTION PROCESS; To reduce the burden of data collectors and make data collection process easier and accessible, data will be collected on google forms/kobo tool. Data collector team will be equipped with android mobile/tab, where kobo tool will be installed. Data will be gathered in offline mode as some of the bordering area, may not have access to internet, once team is back from field will synchronized the data in online mode. This way we will have complete data set at the same time to check quality and completeness, and remove errors through virtual backstopping.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years.
2. Resident of District Haveli, Azad Kashmir for more than last 1 year.
3. Consent to participate in the study.
4. Exposure to war-related stressors (self-reported).

Exclusion Criteria:

1. Age below 18 or above 60 years
2. Ingestion of vit D 200,000 IU in last 3 months.
3. Known diagnosis of primary hyperparathyroidism or sarcoidosis (i.e. conditions pre-disposing to vitamin D hypersensitivity)
4. Residents outside of District Haveli.
5. Baseline corrected serum calcium concentration >2.65 mmol/L
6. Unwillingness to provide informed consent.
7. Medical conditions or medication use affecting vitamin D metabolism.
8. Pregnant or lactating mothers
9. On anti-tuberculosis medicines
10. HIV infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-08-25 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 4 months
  Allostatic load is a measure of physiological dysregulation caused by the accumulated impact of chronic stress on the body.
  Systolic pressure ≥ 150 mmHg, and 120 to 149 mmHg < 120 mmHg Diastolic blood pressure ≥ 90 mmHg, 80 to 89 mmHg < 80 mmHg
lipid profile | 4 months
  Total cholesterol ≥ 240 mg/dL, 200 to 239 mg/dL < 200 mg/dL HDL < 40 mg/dL 40 to 59 mg/dL, > 60 mg/dL Total /HDL cholesterol ≥ 6 5 to < 6 < 5
body mass index BMI | 4 months
  Body mass index (BMI) ≥ 30 kg/m2, and 2 25 to < 30 kg/m2 18 to < 25 kg/m

SECONDARY OUTCOMES:
Serum concentration of vitamin D for the assessment and effect on the allostatic load and chronic stress among the residents of line of control. | 4 months
  Vitamin D level will give us the clue for the supplementation effect and effect on the allostatic load and chronic stress.
  vitamin D normal range 30 ng/dl and above vitamin D insufficiency 20-29 ng/dl vitamin D deficiency less than 20 ng/dl
Hip waist ratio (HRR) cm2 | 4 months
  Waist hip ratio (women) ≥ 0.85cm2 > 0.80 to < 0.85cm2 ≤ 0.80cm2 Waist hip ratio (men) ≥ 1.0cm2 > 0.95 to < 1.0cm2 ≤ 0.95cm2

CONTACTS AND LOCATIONS:
Overall Officials: jawwad AF kayani, PhD, Principal Investigator — University of the Punjab
Locations (1):
- District Headquarter Hospital Haveli, Haveli, Azad Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amrein K, Scherkl M, Hoffmann M, Neuwersch-Sommeregger S, Kostenberger M, Tmava Berisha A, Martucci G, Pilz S, Malle O. Vitamin D deficiency 2.0: an update on the current status worldwide. Eur J Clin Nutr. 2020 Nov;74(11):1498-1513. doi: 10.1038/s41430-020-0558-y. Epub 2020 Jan 20. PMID 31959942
- [Result] Bunting BA, Smith BH, Sutherland SE. The Asheville Project: clinical and economic outcomes of a community-based long-term medication therapy management program for hypertension and dyslipidemia. J Am Pharm Assoc (2003). 2008 Jan-Feb;48(1):23-31. doi: 10.1331/JAPhA.2008.07140. PMID 18192127
- [Result] Casseb GAS, Kaster MP, Rodrigues ALS. Potential Role of Vitamin D for the Management of Depression and Anxiety. CNS Drugs. 2019 Jul;33(7):619-637. doi: 10.1007/s40263-019-00640-4. PMID 31093951